CLINICAL TRIAL: NCT06422260
Title: Clinical and Radiographic Outcomes of Four-unit Implant Supported Fixed Partial Dentures Fabricated From Different Materials
Brief Title: Four-unit Implant Supported Fixed Partial Dentures Fabricated From Different Materials
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, lecturer, Department of prosthodontics, principle investigator, Menoufia University
Other Study IDs: ADMNF-0030324
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Prosthesis Survival; Bone Loss
MeSH Terms: conditions — Prosthesis Failure; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Porcelin fused to metal (PFM) group: Evaluation of biological response and clinical performance of the fixed partial denture anterior bridge constructed from PFM
  Interventions: Other: Prosthesis superstructure
- Zirconia group: Evaluation of biological response and clinical performance of the fixed partial denture anterior bridge constructed from ceramics
  Interventions: Other: Prosthesis superstructure
- Polyetheretherketone (PEEK) group: Evaluation of biological response and clinical performance of the fixed partial denture anterior bridge constructed from PEEK
  Interventions: Other: Prosthesis superstructure

INTERVENTIONS:
Other: Prosthesis superstructure — Prosthesis superstructure for 2 implant supported short span fixed bride constructed from different materials

SUMMARY:
Implant supported superstructure is necessary for long term success and durability of the implant itself in terms of stresses distribution and fracture strength capability. Stresses falling on an implant are too much greater than those applied on a tooth structure with a periodontal ligament offering a degree of elasticity. The important mechanical and physical properties of materials used for the fabrication of dental prostheses include adequate flexural and tensile strength and modulus of elasticity, maximum fracture resistance, optimal bond strength and adequate polishability.

DETAILED DESCRIPTION:
One objective of implant dentistry is to provide excellent esthetics and soft-tissue profiles in the esthetic zone. Esthetic requirements have focused primarily on the position, inclination, shape, and color of the restoration. However, the peri-implant soft tissue also plays a major role in the esthetics of an implant-supported restoration especially in the anterior region.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases that might alter the tissue response to implantation.
* Mobility grade 3 at the site of the 4 lateral incisors.
* sufficient available inter-arch space
* normal maxillomandibular relation.
* no temporomandibular joint

Exclusion Criteria:

* Grade 1 or 2 mobility at the incisor's region.
* Patients with systematic diseases that contraindicate implant placement.

Ages: 30 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: 60 participants who needed an implant-supported fixed partial denture (FPD) in the esthetic zone.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2024-07-22 (Estimated); Study Completion 2025-01-29 (Estimated)

PRIMARY OUTCOMES:
Bone loss | 4 years
  Measurement of alveolar bone loss around implants.

SECONDARY OUTCOMES:
Clinical performance of the prosthesis superstructure | 4 years
  Such as fracture of the prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. El-Sawy, PhD, Principal Investigator — Menoufia University
Locations (1):
- Mohammed A. El-Sawy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
The result can be shared upon request from the corresponding author